CLINICAL TRIAL: NCT02028650
Title: HLA-mismatched Peripheral Hematopoietic Stem Cells Infusion in the Treatment of Leukemia Patients Relapse After HLA- Matched Allogeneic Stem Cell Transplantation: A Randomized Clinical Trial
Brief Title: Randomized Study of HLA-mismatched DSI to Treat Relapse Leukemia After HLA- Matched Transplantation
Status: Completed | Type: Observational
Sponsor: huishengai (Other)
Responsible Party: Sponsor-Investigator, huishengai, director of Hematology Department, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Other Study IDs: RL13-307PLAH-AHS
Record Dates: First submitted 2014-01-01; First posted 2014-01-07 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Relapse Leukemia
Keywords: relapse leukemia; DSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — the blood and bone marrow samples before and after transplantation and DSI
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- the first donor: the original donor applicable patients were assigned to receive the first donor's stem cell treatment after G-CSF mobilization or combination chemotherapy
  Interventions: Biological: the first donor's stem cell
- the second donor: HLA-mismatched, the second donor's stem cell infusion
  Interventions: Biological: the second donor's stem cell

INTERVENTIONS:
Biological: the first donor's stem cell — HLA-matched stem cell infusion
  Groups: the first donor
Biological: the second donor's stem cell — HLA-mismatched, the second donor's stem cell infusion
  Groups: the second donor

SUMMARY:
The relapse leukemia patients after transplantation were divided into two groups randomly. Group D1: patients received first-donor stem cells infusion(DSI) treatment with or without chemotherapy; group D2: patients received second-donor DSI treatment with or without chemotherapy. The second donors were preferably donors who were genetically related and had more HLA-match locus. The re-induction chemotherapy regimen was primarily MAT(mitoxantrone, cytarabine, Teniposide ) for acute myeloid leukemia (AML) and VMCLD(vincristine, Teniposide, cyclophosphamide, L-Asparaginase, Dexamethasone) for acute lymphocytic leukemia (ALL), and no graft versus host disease(GVHD) prevention was conducted pre- and post- therapy.

DETAILED DESCRIPTION:
Evaluation indications include bone marrow morphology,hematopoietic recovery (neutrophil and platelet), 100-day transplantation-related mortality (TRM), donor chimerism, acute GVHD, chronic GVHD, disease free survival (DFS), and overall survival (OS). The cut-time of the follow-up was Oct, 2013. DFS was defined as the time between the date of transplantation to the death or relapse. OS was defined as the time from diagnosis to death or to the last date of follow-up until Oct. 2013.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were between 9 and 67 years of age with de novo diagnosed or treated-related Acute leukemia relapsed after HLA-matched hematological stem cell transplantation from Feb 2005 to Feb 2013
* Relapse was morphologically and molecularly diagnosed,with the help of cytogenetic and engraftment.
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 to 2

Exclusion Criteria:

* Patients without receiving CR will not receive further post-remission trial therapy
* The patients of AML-M3 were excluded from this study.

Ages: 9 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients were between 9 and 67 years of age with de novo diagnosed or treated-related Acute leukemia relapsed after HLA-matched hematological stem cell transplantation from Feb 2005 to Feb 2013.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-02; Primary Completion 2013-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with graft versus host diseases | 100 days

SECONDARY OUTCOMES:
Time to Disease Progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: qiao jianhui, MD, Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality, China